CLINICAL TRIAL: NCT00780559
Title: Improving Neuropathy and Mobility in Subjects With Early Diabetes
Brief Title: Improving Neuropathy and Mobility in People With Early Diabetes
Acronym: INMED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Maryland, College Park (Other); University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B6017-R; INMED 42940 (Other: UMMS IRB)
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-03

CONDITIONS: Diabetes; Physical Activity
Keywords: Neuropathy; diabetes
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity | interventions — Exercise; Standard of Care

STUDY DESIGN:
Intervention Model Description: parallel treatments
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tailored Diet and Physical Activity (Other): Subjects will receive an individually tailored diet and physical activity enhancement program
  Interventions: Behavioral: Tailored Diet and Physical Activity
- Standard of Care (Other): Subjects will be told to reduce their baseline weight by 7% and exercise for 150 minutes/week. There is no tailored, directed program.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Tailored Diet and Physical Activity — Subjects will receive an individually tailored diet and physical activity enhancement program
  Arms: Tailored Diet and Physical Activity
Behavioral: Standard of Care — Subjects will be told to reduce their baseline weight by 7% and exercise for 150 minutes/week. There is no tailored, directed program.
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to determine if an individually tailored diet and physical enhancement program can improve mobility, physical activity, and neuropathy in people with early diabetes.

DETAILED DESCRIPTION:
Neuropathy is the most common complication of diabetes mellitus. Impaired glucose regulation (IGR) is associated with development of peripheral neuropathy coupled with gait and mobility impairment that may be disabling for the patient. Recent novel data from the investigators' group indicates that improved diet and exercise can significantly improve and even reverse neuropathy associated with IGR, however this has not been tested as a specific intervention in a controlled diabetes complications trial. IGR includes patients with early type 2 diabetes mellitus (T2DM), impaired glucose tolerance (IGT), and impaired fasting glucose (IFG) based on standardized criteria for the diagnosis of T2DM. The investigators hypothesize that, compared to IGR participants advised to follow the current standard care recommendations on diet and exercise (Standard Care or "SC"), IGR participants undergoing a Tailored Diet and Physical Activity (TDPA) enhancement program will show greater improvement in the 6 minute walk test (6MW) and will show a greater reduction in markers of neuropathy progression e.g. intraepidermal nerve fiber density (IEFND). Furthermore, the investigators will test the hypothesis that improvement in measures of neuropathy, mobility function and physical activity (PA) will correlate strongly with each other and with improvement in specific measures of metabolic function, and weight loss. This proposal will permit us to determine if TDPA can improve mobility and induce nerve regeneration in subjects with early diabetes.

ELIGIBILITY:
Inclusion Criteria:

* IGR at the time of screening or within three months of screening. This definition includes patients with impaired fasting glucose (IFG), impaired glucose tolerance (IGT), and early diabetes. Patients can be included if they have an increased risk for diabetes with a HBA1C > or = 5.7% (using a method certified by the National Glycohemoglobin Standardization Program), or they have diabetes with a HBA1C > or equal to 6.5%, or an abnormal fasting venous glucose, or abnormal venous glucose values following a 75 gram oral load. Glucose values are as defined (mg/dl): IFG fasting greater than 100 mg/dl, IGT- fasting less than 126, 2 h 140-199, or diabetes - fasting glucose > 126, 2 h > 200 based on the Standards for Medical Care in Diabetes 2010 by the American Diabetes Association.
* The HbA1c may be normal, but must be <8%.
* If diabetic subjects are on medication, they should be stable on medication for at least 3 months prior to entering the study. Addition or change in antidiabetic medications after enrollment does not affect participation or group assignment.
* No risk factors for other causes for neuropathy (determined by a medical history, family history, history of medications, occupational history, history of exposure to toxins, physical and neurological examinations, and laboratory studies).
* Clinical signs or symptoms of neuropathy as determined by the treating neurologists history and physical exam, plus an abnormality of one of the following: nerve conduction studies (NCS), Quantitative Sudomotor Autonomic Reflex Testing (QSART), Quantitative Sensory Testing (QST), or IENFD.
* Age range from 30 to 80 years inclusive at the time of screening
* Medically stable at the time of enrollment.
* Able to participate in a standing exercise program without constant standby monitoring.
* Women of childbearing potential must be using an acceptable method of contraception to prevent pregnancy when they are enrolled in the study and must agree to continue to practice an acceptable method of contraception for the duration of their participation in the study.
* Patient must agree to taking an alternative medication to coumadin when undergoing a skin biopsy
* Willing to complete weekly self-report questionnaires.
* Willing to accept assignment to either training group.
* Willing and able to increase activity level and exercise independently at home.

Exclusion Criteria:

* Pregnant women, prisoners, institutionalized subjects and other at risk subjects will not be included in this study.
* Taking insulin.
* Etiology of sensorimotor neuropathy other than IGR based on careful clinical and laboratory evaluation.
* Current severe medical conditions that are active on the day of enrollment and would affect a patient's ability to complete study. This may include active advanced current ischemic heart disease (e.g., angina or congestive heart failure), permanent residual lower extremity weakness or loss of balance resulting from a stroke, active severe obstructive or restrictive pulmonary disease, ongoing cancer treatment, renal failure currently requiring dialysis, or severe ongoing peripheral vascular disease.
* An inability to understand or cooperate with the procedures of the trial or refusal to sign the informed consent.
* Patients who are unable to answer questions correctly on the Evaluation to Sign Consent (ESC) tool.
* Significant other neurologic, rheumatological, neuromuscular, or other extremity conditions that limit safe exercise or weight bearing.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-11-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James W Russell, MD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (3):
- United States (3):
  - University of Maryland, Baltimore, Maryland
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were excluded from the study prior to assignment for groups (n=12) due to failure of screening (e.g. not meeting inclusion/exclusion criteria, n=10) or declined to participate (n=2.)
Period: Overall Study
Arm/Group | Tailored Diet and Physical Activity | Standard of Care
Started | 32 | 40
Completed | 29 | 33
Not Completed | 3 | 7
Not completed — Lost to Follow-up | 2 | 7
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants were IGR patients with neuropathy, including early type 2 diabetes mellitus (T2DM - within 2 years of diagnosis), impaired glucose tolerance (IGT), and impaired fasting glucose (IFG) patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tailored Diet and Physical Activity | Standard of Care | Total
Number analyzed (Participants) | 32 | 40 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 28 | 46
  >=65 years | 14 | 12 | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.81 (8.25) | 61.03 (7.83) | 61.38 (7.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 21 | 27 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 7 | 12
  White | 26 | 30 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
BMI (Body Mass Index), Categorical [Count of Participants; unit: Participants] — Body Mass Index defined as kg/m^2 at the time of screening/baseline visit.
  Participants
    BMI < 30 kg/m^2 | 13 | 19 | 32
    BMI 30 - 40 kg/m^2 | 12 | 19 | 31
    BMI > 40 kg/m^2 | 7 | 2 | 9
BMI (Body Mass Index), Continuous [Mean (Standard Deviation); unit: kg/m^2] | 33.21 (7.65) | 30.83 (7.06) | 31.89 (7.37)

OUTCOME MEASURES:

1. Primary Outcome: Six Minute Walk (6MW) Test
Description: Measures distance covered by participant when walking at a brisk pace without running for six minutes in feet.
Time Frame: Six Months
Measure: Least Squares Mean (Standard Error); unit: feet
Arm/Group | Tailored Diet and Physical Activity | Standard of Care
Number analyzed (Participants) | 32 | 40
feet | 156.644156 (35.364227) | 61.257846 (35.840649)

2. Primary Outcome: Change in 6-Minute-Walk Test Measured in Feet Between Baseline and 12 Months
Time Frame: Baseline and 12 Months
Measure: Least Squares Mean (Standard Error); unit: feet
Arm/Group | Tailored Diet and Physical Activity | Standard of Care
Number analyzed (Participants) | 32 | 40
feet | 188.415845 (34.346235) | 100.559319 (36.399507)

3. Secondary Outcome: Intraepidermal Nerve Fiber Density (Distal Leg)
Description: Measure of the number of skin fibers/mm in the lower extremity (distal leg) at 12 months
Time Frame: 12 Months
Measure: Least Squares Mean (Standard Error); unit: fibers/mm
Arm/Group | Tailored Diet and Physical Activity | Standard of Care
Number analyzed (Participants) | 32 | 40
fibers/mm | 1.28627099 (0.81830712) | -0.38943425 (0.84781677)

4. Secondary Outcome: Intraepidermal Nerve Fiber Density (IENFD) at the Proximal Thigh
Description: Measure of the number of skin fibers/mm in the lower extremity (proximal thigh) at 12 months
Time Frame: 12 Months
Measure: Least Squares Mean (Standard Error); unit: fibers/mm
Arm/Group | Tailored Diet and Physical Activity | Standard of Care
Number analyzed (Participants) | 32 | 40
fibers/mm | 1.53825016 (0.83395303) | -0.54419990 (0.87926529)

5. Other Pre Specified Outcome: Change in Physical Activity (PA) at 12 Months as Measured by the CHAMPS (Community Health Activities Model Program for Seniors) Activity Scale
Description: Physical Activity measured by CHAMPS provides an estimated caloric expenditure of subject based on weight and weekly physical activity, as assessed by the questionnaire. Change in physical activity is determined by the difference in daily caloric expenditure at baseline and 12 months.
Time Frame: Baseline and 12 Months
Measure: Least Squares Mean (Standard Error); unit: kcal/day
Arm/Group | Tailored Diet and Physical Activity | Standard of Care
Number analyzed (Participants) | 32 | 40
kcal/day | -735.249060 (886.986000) | 296.998122 (937.935990)

ADVERSE EVENTS:
Time Frame: Adverse event data for each participant was collected over one year per study patient, or the duration of the study for each participant.
Description: The definition of adverse events and/or serious adverse events does not differ from that which is listed here on clinicaltrials.gov. Adverse Events were collected from patient reports and phone call follow-ups.
Arm/Group | Tailored Diet and Physical Activity | Standard of Care
All-Cause Mortality (participants affected / at risk) | 1/32 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/40
Other Adverse Events (participants affected / at risk) | 1/32 | 0/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tailored Diet and Physical Activity (N=32) | Standard of Care (N=40)
Skin Irritation (Product Issues) | 1 (1) | 0 (0) — Participant complained of skin rash at biopsy wound site. This is not outside of risks, and participant was irritated by the bandage.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-09-09): https://cdn.clinicaltrials.gov/large-docs/59/NCT00780559/Prot_SAP_000.pdf